CLINICAL TRIAL: NCT06533072
Title: The Effect Of Infrared Led Lıght Applıcatıon On Wound Healıng, Scar And Scar Tıssue Formatıon In Patıents Havıng Laparascopıc Cholesystectomy Surgery
Brief Title: Infrared LED Lighting Application and Wound Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Responsible Party: Principal Investigator, Gülistan UYMAZ ARAS, lecturer, Ardahan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: arasuymazgulistan
Record Dates: First submitted 2024-07-22; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cholecystectasia; Wound Heal; Scar
Keywords: surgical wound; Photobiomodülation; Ligh; Therapy
MeSH Terms: conditions — Cicatrix; Surgical Wound

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients who received routine medical treatment and nursing care + IR LED Light application after surgery (n = 40). It is applied on Post-Operative Day 1-2. It will be given four times in total, from a distance of 45-60 cm, for 20 minutes at 8 hour intervals (Wolters and Feaarnly, 2023). The patient will be asked to remain in the supine position during the procedure and the patient's vital signs will be checked again after the procedure. After the third and last Infrared LED application on post-op Day 2, the patient's wound was re-evaluated and the wound was dressed and closed. On the 15th and 30th post-operative day, the patient will be asked to come to the hospital and the wound site will be re-evaluated and the data collection form will be filled out again.
  Interventions: Other: The group receiving infrared LED therapy
- Control group (No Intervention): This is the group of patients who received routine medical treatment and nursing care after surgery (n=40). After the patient's vital signs were taken postoperative one day and after the Informed Consent Form was obtained from patients who met the inclusion criteria and volunteered to participate in the study; Data collection form (demographic information form, Bates-Jensen wound assessment scale, observer scar assessment scale, VAS, Newcastle Nursing Care Satisfaction Scale) will be filled out.

INTERVENTIONS:
Other: The group receiving infrared LED therapy — Patients in this group are the ones who will be exposed to IR LED light therapy, three times in total
  Other Names: experimental group
  Arms: experimental group

SUMMARY:
Laparoscopic cholecystectomy is a commonly used procedural procedure for removal of the gallbladder. Following this healing, wound healing, scar formation and scar tissue formation are critical factors in the healing process. The development of painless, noninvasive, biophysical therapeutic interventions has become the focus of current biomedical research. In recent years, it has been reported that infrared (IR) LED light applications have positive effects on tissue healing processes. This study will be conducted in a randomized controlled manner to examine the effect of postoperative IR LED application on wound healing, scarring and scar tissue formation in patients who underwent laparoscopic cholecystectomy.The research will be carried out at Erzurum City Hospital General Surgery Clinic between 15.08.2024-30.08.2025. A number sequence will be created for the 80 patients in the sample who meet the inclusion criteria for the experimental group and control group, and they will be assigned to the experimental (n = 40) and control groups (n = 40) using a computerized randomization program (https://www.random.org/integer-sets/) patient distribution will be provided. First of all, IR LED light application; It is applied on Post-Operative Day 1 and postoperative day 2. It will be given four times in total, from a distance of 45-60 cm, for 20 minutes at 8 hour intervals. On the 15th and 30th post-operative day, the patient will be asked to come to the hospital and the wound site will be re-evaluated and the data collection form will be filled out again. The patient's pain status will be evaluated with VAS, and satisfaction with Newcastle Nursing Care Satisfaction Scale. Wound and scar tissue will be examined with the Bates Jensen wound assessment scale and the patient and observer scar assessment scale. Wound and scar sites will be re-evaluated after the 15th and 30th post-operative day. The patient's pain status will be evaluated with VAS, and satisfaction with Newcastle Nursing Care Satisfaction Scale. Wound and scar tissue will be examined with the Bates Jensen wound assessment scale and the patient and observer scar assessment scale. The wound margin will be measured with a disposable ruler. In coding and evaluating the data; SPSS 22.00 package program will be used.

DETAILED DESCRIPTION:
1. Introduction Laparoscopic cholecystectomy is a commonly used procedural procedure for removal of the gallbladder. Following this healing, wound healing, scar formation and scar tissue formation are critical factors in the healing process. There are countless wounds; The development of painless, noninvasive, biophysical therapeutic interventions has become the focus of current biomedical research. In recent years, it has been reported that infrared (IR) LED light applications have positive effects on tissue healing processes. IR LED red light application has recently become a widely preferred method due to its ease of application, easy access, no need for expertise for application, and the ability of individuals to apply it at home or anywhere they want. The ability of light to penetrate a tissue and accumulate energy through the tissue's optical absorption properties is key to therapeutic applications. When electromagnetic radiation strikes biological tissue, different interactions occur as a function of various physical parameters. In the medical field, red and near-light induced IR LED (Low Energy Light) application (therapy) is known for its abilities to promote wound healing, reduce inflammation, reduce pain, and positively modulate biochemical and molecular chemicals. Although the light-tissue interaction depends primarily on wavelength, it is also affected by the tissue components that interact with the photons. In tissue, an 'optical window' lies between 600 and 1350 nm. Light with a wavelength smaller or larger than this region is absorbed by tissue components (hemoglobin, myoglobin in the visible region and tissue water content in the IR region). Additionally, biological tissue has a lower scattering capacity in the NIR region than in the visible region. This means that biological experiments in this range can be performed without damaging skin tissue. This has led to the emergence of new hopes for the destruction of microorganisms on the skin before they develop resistance, providing painless treatment with light-based treatments, and chronic wound healing. Although the wound area is minimal in patients who undergo cholecystectomy by laparoscopy method, the healing time of the wound varies between 3 weeks and 8 weeks and this period may be longer depending on the condition of the individual. The location of the wound in the abdomen restricts the patient's movements and leaves a scar in the abdomen. This situation negatively affects the patient psychologically and socially. In the study, patients who underwent minimally invasive surgery were selected because they provide a better opportunity to observe the wound site, as external factors can be more easily controlled, the hospitalization period, infection and other physical complications are less likely. Therefore, the smaller the wound area, the easier the wound can be closed and the scar can be seen more quickly, making it easier to work. In patients who undergo surgery with minimal laparoscopy, the postoperative care protocol is more focused on medical treatment and long-term effects are ignored. Our study offers a different postoperative care protocol for patients undergoing minimally invasive surgery. There is no certainty in the literature regarding the duration and intervals of LED application to the wound site. Kim et all applied light with 660 wavelengths at different distances to the wound site once and reported that application for 10 minutes better increased the activity at the cell level. In a different study, it was found that two applications were made instead of the incision after cesarean section surgery, but no clear information was found in the study about the number of hours between applications. In the study, the wound site was evaluated on the 3rd day before the patient was discharged. In a case report reported by Vinck et all a male patient who had an operation on his foot applied light at a wavelength of 950 nm to the 6 cm incision. The evaluation was made 6 days later. It was reported that there was less color change and less scarring in the 2.6 cm area. It is planned to perform a control evaluation on the 15th and 30th days post-op to compare the thickness of the scar tissue and the change in the wound site. During the research process, patients' wound healing will be observed, scar formation will be evaluated, and scar tissue formation will be examined. Various ancillary parameters will also be recorded, including patient satisfaction, pain levels, and other factors in the healing process. The results of this research will reveal the potential effects of IR LED light application on wound healing, scar formation, and scar tissue formation after laparoscopic cholecystectomy. These findings are important for developing new treatment strategies to optimize post-surgical recovery processes. The findings may offer clinicians new perspectives on optimizing patient care after surgical intervention. The following hypotheses will be tested in the research.

Ho: Application of IR LED light to the wound site has no effect on wound healing.

H1: Application of IR LED light to the wound site has a positive effect on wound healing.

Methods Type of Research This study will be conducted in a randomized controlled manner to examine the effect of postoperative IR LED application on wound healing, scarring and scar tissue formation in patients who underwent laparoscopic cholecystectomy.

Place and Time of Research The research will be carried out at Erzurum City Hospital General Surgery Clinic between 30.06.2024-30.08.2025.

Universe of Research The population of this research will consist of patients who underwent surgery with Laparoscopic Cholecystectomy at Erzurum City Hospital between June 2024 and August 2025.

Sample of the Research In order to examine wound healing, scarring and scar tissue formation in patients undergoing laparoscopic cholecystectomy surgery, the sample size of the study was; Calculated using G*Power statistical program (ver.3.1.9.7)*. According to this; Taking Power 0.95, Effect size 0.4034733 (Eta squared 0.14) and Type-1 error (a) 0.05 (for control and experimental groups), the number of patients was determined as 66 patients, with a minimum of 33 (sample) in each group. However, due to possible data loss, 10-20% was added to the sample number and 40 patients were determined for each of the experimental-control groups, 80 patients in total. A number sequence will be created for the 80 patients in the sample who meet the inclusion criteria for the experimental group and control group, and they will be assigned to the experimental (n = 40) and control groups (n = 40) using a computerized randomization program (https://www.random.org/integer-sets/) patient distribution will be provided. Before starting the research, a preliminary application will be made at Erzurum City Hospital with 10 patients (5 experimental and 5 control) who underwent laparoscopic cholecystectomy. Work will begin after preliminary application.

Criteria for inclusion in the study 1.Being 18 years or older, 2. Being 65 years old 3. Volunteer to participate in the study 4. Having cognitive competence 5. Absence of any chronic disease (diabetes, COPD, hypertension, etc.) 6. Not Separating the Wound 7. Tympanic body temperature; 35.7-37.5; axillary; It should be between 36.5 and 37.0 Study exclusion criteria 1. Presence of signs and symptoms of infection at the wound site 2. Unusual bleeding at the wound site 3. Patients are given hypertensive, anticoagulant, thyroid etc. starting medications Data Collection Tools In order to be applied to the experimental group, an infrared device, a patient introduction form created in line with the literature as a data collection tool, a wound measurement ruler, a Bates-Jensen wound evaluation tool, a patient and observer scar evaluation scale, a visual analogue scale (VAS) to question the pain level, and a Newcastle scale to question the satisfaction level were used. Nursing Care Satisfaction Scale (NHBMS) will be used.

1. Patient Introduction Form This form, prepared by the researchers, consists of a total of 17 questions to inquire about the socio-demographic characteristics of the patients and their disease-related characteristics.
2. Wound Measuring Ruler Wound measuring ruler is a measuring tool used in hospitals and health centers. This ruler is used to measure the size, depth and other characteristics of wounds. Wound measuring rulers can come in various shapes and sizes, usually in the form of post-it notes.
3. Bates-jensen Wound Assessment Tool The assessment tool developed by Bates-Jensen et al. in 1992 is a scale that broadly considers the physiological and anatomical features of the wound. It consists of 13 items: size, depth, edges, tunneling, type and amount of necrotic tissue, type and amount of exudate, color of the skin around the wound, peripheral tissue edema and hardness around the wound, granulation tissue and epithelialization. As a result of the scale scoring, 1 point indicates that the wound is in better condition, and 5 points indicates that the wound condition is worse. In the presence of necrotic tissue, the type and amount of necrosis are also included in the evaluation. The total score obtained varies between 13-65, and an increase in the score indicates that the wound condition is worsening.
4. Patient and Observer Scar Evaluation Scale The Patient and Observer Scar Assessment Scale was developed by Draaijers et all. (2004) in 2004 to evaluate burn wounds. Although the validity and reliability of the scale was conducted on burn wounds, it is seen that it is used for scar evaluation in surgical wounds and it is stated that the scale can be used for scar evaluation of surgical wounds The quality of the scar is characterized by the presence or absence of certain features by looking, touching and feeling. Basically, the scar is evaluated by its color, surface texture, flexibility, thickness, surface area, pain and itching characteristics. The scale consists of a total of 7 items, 6 of which are used to evaluate the scar (evaluation of pain, itching, color, flexibility, thickness and irregularity) and 1 of which evaluates the general opinion about the scar. Each item has a Likert type scoring between 1 and 10. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get from the scale is 6, which indicates normal skin, and the highest score, 60, represents the worst scar imaginable, and the scale score is calculated based on the first 6 items. The 7th article, which questions the general opinion about scars, has only a scoring criterion and is evaluated among itself. In determining scar tissue thickness; average distance between the subcutaneous-dermal border and the epidermal surface of the scar; The scar will be evaluated by touching it with the fingertips. It will be decided whether the scar tissue is thin or thick, taking into account its difference from the epithelial tissue, its strength and hardness, and it will be marked as thin or thick on the scale. To evaluate pigmentation; Plexiglass is placed on the wound with moderate pressure and scored by comparing it with the pigmentation of intact skin. To evaluate vascularization, plexiglass is placed on the wound and the color of the wound is pale by applying pressure, then the plexiglass is removed and the vascularization of the wound is observed. When assessing wound site irregularity, the extent of existing surface irregularities is compared with adjacent normal skin. As a result of the comparison, it is checked whether the scar tissue is puffier than normal tissue. The elasticity of the scar is evaluated by squeezing the scar between the thumb and index finger. When evaluating the surface area, the tendency for the scar to grow or shrink compared to the initial time will be evaluated. Photography technique is used to determine whether there is expansion or contraction in the surface area of the scar.
5. Visual Analog Scale (VAS) It is a scale used to convert some values that cannot be measured numerically into numerical values. The scale consists of numbers from 1 to 10 placed one centimeter apart on a 10-centimeter horizontal ruler. The scale is a pain assessment tool that has proven itself for a long time and is accepted in the world literature.
6. Newcastle Nursing Care Satisfaction Scale (NNCSS) The scale was developed by Thomas and Bond in 1996, adapted to Turkish by Uzun in 2003, and Akın and Erdoğan in 2007, and its validity and reliability studies were conducted. It is a 19-item, single-subdimensional, five-grade Likert-type scale. All items of the scale take values between 1 and 5, and the values of all marked items are summed and converted to 100. Total score evaluation is made on a scale of 0-100. A total score close to 100 indicates satisfaction with nursing care. The Cronbach internal consistency coefficient of the scale was found to be 0.96 in the study of Thomas et all.

Enterprise Materials 1. Infrared Device: The device is a treatment device that uses light currents and has a system that can cause moderate or strong therapeutic effects on the body area and surface with the light and heat it emits. It is used for regional treatment by utilizing infrared light and adjusting the wavelengths according to the areas suitable for the treatment area, thus heating that area. The device has the ability to emit adjustable red light at 630-700 wavelengths.

Collection of Data

1. Data Collection from Experimental Group Patients

1. Patients who received routine medical treatment and nursing care + IR LED Light application after surgery (n = 40).
2. Post-op 1. day; After taking the patient's vital signs between hours, the 'Informed Volunteer Consent Form' was obtained from patients who met the inclusion criteria and volunteered to participate in the study; Before IR LED application, a data collection form (patient introduction form, Bates-Jensen scar evaluation scale, patient and observer scar evaluation scale, VAS, Newcastle Nursing Care Satisfaction Scale) will be filled out. A disposable wound measurement ruler, Bates Jensen wound evaluation scale, and Observer Scar Evaluation Scale will be used to evaluate the wound site. Images will be taken with a DSLR camera to be used to evaluate the wound scar surface area.
3. First of all, IR LED light application; It will be given four times in total, from a distance of 45-60 cm, for 20 minutes at 8 hour intervals. The patient will be asked to remain in the supine position during the procedure and the patient's vital signs will be checked again after the procedure. The critical time for wound healing is the first 24-72 hours after surgery. After the third and last IR LED application on post-op Day 1, the patient's wound was re-evaluated and the wound was dressed and closed.
4. Scar development begins to become evident on the 14th day following wound formation. On the 15th and 30th post-operative day, the patient will be asked to come to the hospital and the wound site will be re-evaluated and the data collection form will be filled out again. The patient's pain status will be evaluated with VAS, and satisfaction with Newcastle Nursing Care Satisfaction Scale. Wound and scar tissue will be examined with the Bates Jensen wound assessment scale and the patient and observer scar assessment scale. The patient will also be asked to complete the Patient and Observer Scar Assessment Scale, the Patient Scar Assessment Scale, to assess his or her scar status.
5. In evaluating the wound boundaries, the measurement of the wound will be made using a disposable wound measurement ruler and the measurement of the wound will be recorded on the data collection form. Scar evaluation will be made with the "Patient and Observer Scar Evaluation Scale". To evaluate the thickness, the average distance between the subcutaneous-dermal border and the epidermal surface of the scar; The scar will be evaluated by touching it with the fingertips. It will be decided whether the scar tissue is thin or thick, taking into account its difference from epithelial tissue, its strength and hardness.

1. Data Collection from Control Group Patients

1. This is the group of patients who received routine medical treatment and nursing care after surgery (n=40).

6. After the patient's vital signs; the Informed Volunteer Form was obtained from patients who met the inclusion criteria and volunteered to participate in the study; Data collection form (demographic information form, Bates-Jensen wound assessment scale, observer scar assessment scale, VAS, Newcastle Nursing Care Satisfaction Scale) will be filled out. A disposable wound measurement ruler, Bates Jensen wound evaluation scale, and Observer Scar Evaluation Scale will be used to evaluate the wound site. Images will be taken with a DSLR camera to be used to evaluate the wound scar surface area.

7. After the 15th and 30th post-operative day, the patient will be asked to come to the hospital and the wound site will be re-evaluated and the data collection form will be filled out again. The patient's pain status will be evaluated with VAS, and satisfaction with Newcastle Nursing Care Satisfaction Scale. Wound and scar tissue will be examined with the Bates Jensen wound assessment scale and the observer scar assessment scale. The wound border will be measured with a disposable ruler.

8. In evaluating the wound boundaries, the measurement of the wound will be made using a disposable wound measurement ruler and the measurement of the wound will be recorded on the data collection form. Scar evaluation will be made with the "Patient and Observer Scar Evaluation Scale". To evaluate the thickness, the average distance between the subcutaneous-dermal border and the epidermal surface of the scar; The scar will be evaluated by touching it with the fingertips. It will be decided whether the scar tissue is thin or thick, taking into account its difference from epithelial tissue, its strength and hardness.

Analysis of Data In evaluating the data; In addition to standard deviation, mean, number and percentages, it is thought that analyzes such as t-test in independent groups, t-test in dependent groups, analysis of variance, correlation and regression analysis will be used in statistical comparisons, depending on the characteristics of the data. Normal distributions of the data will be evaluated using Kurtosis and Skewness coefficients, and non-parametric tests will be used for data that do not show normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years and under 65 years old
* Volunteer to participate in the study
* Having cognitive competence
* Absence of any chronic disease (diabetes, COPD, hypertension, etc.)
* Not Separating the Wound
* Tympanic body temperature; 35.7-37.5; axillary; It should be between 36.5 and 37.0

Exclusion Criteria:

* Presence of signs and symptoms of infection at the wound site
* Unusual bleeding at the wound site
* Patients are given hypertensive, anticoagulant, thyroid etc. starting medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
wound healing | 1 month
  To accelerate wound healing with postoperative infrared LED light application
Scar Tıssue Formatıon | one month
  scars can create functional problems for patients. It is aimed to provide a more cosmetic and aesthetic appearance by preventing scar formation.

SECONDARY OUTCOMES:
physiological parameter | one month
  Increasing patient satisfaction not only affects recovery but also strengthens communication between healthcare professionals and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karaman Özlü, PhD, Study Director — Atatürk Universty
Locations (1):
- Atatürk Universty, Erzurum, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No